CLINICAL TRIAL: NCT02781389
Title: Non-interventional Study to Investigate the Effectiveness, Safety and Utilization of Vismodegib on Locally Advanced Basal Cell Carcinoma Under Real World Conditions
Brief Title: Vismodegib on Locally Advanced Basal Cell Carcinoma Under Real World Conditions
Acronym: JONAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: OnkoDataMed GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Dirk Schadendorf, Prof. Dr. med., University Hospital, Essen
Other Study IDs: ML29828
Record Dates: First submitted 2016-04-24; First posted 2016-05-24 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma (BCC); advanced BCC (aBCC)
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this non-interventional study is to provide further data on the utilization, effectiveness, safety and clinical benefit including duration of response of Vismodegib for treatment of locally advanced basal cell carcinoma (laBCC), inappropriate for surgery or radiotherapy under real world clinical conditions.

DETAILED DESCRIPTION:
This is a multi-center non-interventional study with 53 patients with locally advanced BCC who start Vismodegib (received at least one dose) in Q4 2015. Duration of recruitment will be one year. Patients will be followed prospectively until disease progression, death, or for 3 years from first dose Vismodegib (whichever occurs first).

The primary effectiveness objective for this study is as follows:

• To evaluate the duration of response defined as duration from first documented response of complete response (CR) or partial response (PR) until disease progression (as determined by the treating physician, which might include and will be categorized in the following groups: clinical assessment, histological assessment, imaging assessment) for laBCC patients.

The secondary effectiveness objectives for this study are as follows:

* Objective response rate (rate of patients with CR or PR) (as determined by the treating physician, which might include and will be categorized in the following groups: clinical assessment, histological assessment, imaging assessment)
* Disease control rate (complete response (CR), partial response (PR) or stable disease (SD))
* Recurrence rate: rate of patients who responded (CR or PR) and later progressed
* Time to progression: time from first treatment to progression
* Time to death: time from first treatment to death
* Time to response: time from first treatment to response

The explorative objectives of this study are to evaluate the following endpoints:

* Type of tumor response evaluation (as determined by the treating physician, which might include and will be categorized in the following groups: clinical assessment , histological assessment, imaging assessment)
* Treatment decision for therapy with Vismodegib (tumor board OR decision by otorhinolaryngologist, surgeon, plastic surgeon, dermato-oncologist, radiotherapist, ophthalmologist)
* Utilization

  * Previous treatment for the BCC lesion, which led to therapy with Vismodegib
  * BCC therapy after Vismodegib therapy (if applicable)
  * Treatment duration of Vismodegib (start and stop dates for therapy with Vismodegib)
  * Assessment of duration and time point of treatment interruptions of Vismodegib
  * Reason for treatment discontinuation

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age ≥ 18 years
* laBCC (inappropriate for surgery or radiotherapy)
* Patient is not included in any other trial
* Male or female patient is included in the pregnancy prevention program, as determined by the German authority (BfArM)

Exclusion Criteria:

Patients, for whom treatment with Vismodegib is contraindicated according to the Summary of Product Characteristics (SmPC), which has been in effect at the time of treatment with Vismodegib, including:

* Hypersensitivity to the active substance or to any of the excipients listed in section 6.1. of the latest SmPC
* Women who are pregnant or breast-feeding
* Women of childbearing potential who do not comply with the Vismodegib (Erivedge) Pregnancy Prevention Programme
* Coadministration of St John's wort (Hypericum perforatum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 53 Patients with locally advanced BCC who are being treated with Vismodegib will be followed prospectively by centers across Germany and clinical course will be documented
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Primary effectiveness measure: duration of response (partial or complete) until progression, death or up to 3 years from first dose Vismodegib (whichever occurs first) | up to 3 years from first dose Vismodegib
  The primary effectiveness measure for this study is as follows:
  • To evaluate the duration of response, defined as duration from first documented complete response (CR) or first documented partial response (PR), whichever cam first, until disease progression (as determined by the treating physician), or death of any reason or up to 3 years from first dose Vismodegib, whichever occurs first, for laBCC patients.

SECONDARY OUTCOMES:
Secondary effectiveness measure: - objective response rate | up to 3 years from first dose Vismodegib
  number of patients with complete response or partial response as determined by the treating physician by clinical assessment, histological assessment, imaging assessment
Secondary effectiveness measure: - time to response | up to 3 years from first dose Vismodegib
  time from first dose Vismodegib to complete response or partial response up to 3 years
Secondary effectiveness measure: - disease control rate | up to 3 years from first dose Vismodegib
  number of complete response, partial response, stable disease
Secondary effectiveness measure: - recurrence rate | up to 3 years from first dose Vismodegib
  number of patients who responded (partial or complete) and later progressed
Secondary effectiveness measure: - time to progression | up to 3 years from first dose Vismodegib
  time from first dose Vismodegib to progression up to 3 years
Secondary effectiveness measure: - survival | up to 3 years from first dose Vismodegib
  time from first dose Vismodegib to death of any cause

OTHER OUTCOMES:
Explorative outcome measures: tumor response | up to 3 years from first dose Vismodegib
  - type of tumor response as determined by the treating physician by clinical assessment and/or histological assessment and/or imaging assessment
Explorative outcome measures: treatment decision for therapy with Vismodegib | up to 3 years from first dose Vismodegib
  - treatment decision for therapy with Vismodegib by tumor board OR by otorhinolaryngologist, surgeon, plastic surgeon, dermato-oncologist, radiotherapist, ophthalmologist
Explorative outcome measures: previous treatment | up to 3 years from first dose Vismodegib
  - previous treatment for the BCC lesion, which led to therapy with Vismodegib
Explorative outcome measures: therapy after Vismodegib | up to 3 years from first dose Vismodegib
  - BCC therapy after Vismodegib therapy
Explorative outcome measures: duration of therapy with Vismodegib | up to 3 years from first dose Vismodegib
  - time of treatment with Vismodegib
Explorative outcome measures: Vismodegib therapy interruptions | up to 3 years from first dose Vismodegib
  - time to treatment interruptions of Vismodegib
Explorative outcome measures: Vismodegib treatment discontinuation | up to 3 years from first dose Vismodegib
  - reason for treatment discontinuation of Vismodegib

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Professor, Principal Investigator — Universitätsklinikum Essen
Locations (1):
- Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie (Universitätsklinikum Essen), Essen, Germany

IPD SHARING:
Plan to Share IPD: No